CLINICAL TRIAL: NCT06185439
Title: The Effect of Prenatal Pilates-Supported Childbirth Training on Birth Outcomes and Incontinence: A Randomized Controlled Study
Brief Title: Prenatal Pilates Assisted Childbirth Preparation Training and Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gonca Buran, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-KAEK-26/193
Record Dates: First submitted 2023-12-05; First posted 2023-12-29 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Incontinence, Urinary; Training Group, Sensitivity
Keywords: Pregnancy pilates; Urinary incontinence; childbirth training
MeSH Terms: conditions — Urinary Incontinence; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Following recruitment, the pregnant women were divided into a study and a control group by randomization (1:1 randomization)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The data will be collected by the assistant researcher and entered into the SPSS program as A and B groups. Analyzes will be performed by the principal investigator who is blind to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Study group (Experimental): In this study, the study group was provided with prenatal pilates-assisted childbirth preparation training and follow-up, in addition to the usual care provided by health professionals.
  Interventions: Behavioral: Prenatal Pilates Assisted Childbirth Preparation Training
- Control group (No Intervention): The control group was in the usual care.

INTERVENTIONS:
Behavioral: Prenatal Pilates Assisted Childbirth Preparation Training — Training was given twice a week for two hours a day (one hour of theory, one An hour of exercise = 45 minutes of pregnant plates and 15 minutes of breathing exercises) total eight weeks.
  Other Names: Experimental: Study group
  Arms: Experimental: Study group

SUMMARY:
A randomized controlled trial was made to determine the effectiveness of prenatal pilates-supported childbirth preparation training on birth outcomes, incontinence during pregnancy, and the postpartum period.

DETAILED DESCRIPTION:
One of the risk factors for the development of stress incontinence in women is pregnancy and childbirth. This problem increases as pregnancy progresses and continues in the postpartum period.

It was tested the hypothesis, there is no difference in the development of urinary incontinence in the prenatal and postpartum periods among women who receive Pilates-assisted childbirth preparation training and women who were into the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35,
* Being in the 28th-30th week of pregnancy
* Having a singleton pregnancy
* Being nulliparous

Exclusion Criteria:

* Having chronic constipation
* Having a chronic cough
* Having a history of any psychiatric condition, multiple sclerosis, spinal cord injury, congenital or acquired anatomical abnormalities of the urogenital tract, bladder malignancy
* Being overweight and obese
* Giving birth outside of 37-42 weeks

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — for pregnancy
Enrollment: 126 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Pre-intervention | During assessment at registration
  During the prenatal period, evaluation of incontinence score with the Michigan Incontinence Severity Index Form (minimum score : 0- maximum score:40) during an assessment at registration before intervention (before education and pilates). A score higher than the given cut-off values indicates that the severity of incontinence is worsening.
Intervention- Childbirth training program and prenatal pilates intervention | Immediately after at the end of the eight-week prenatal pilates-supported birth preparation training
  Evaluation of incontinence score with the Michigan Incontinence Severity Index Form ( minimum score: 0 -maximum score: 40 cut of the point: 7 and above ) after the intervention. Questions 1st-3th on the MISIF scale indicate stress incontinence severity, 4th-6th questions measure the severity of urge incontinence, and 1st-8th questions measure the severity of incontinence. There points above indicate stress incontinence and the total score of questions 4-6 indicates 5 points and above for urge incontinence severity.A score higher than the given cut-off values indicates that the severity of incontinence is worsening.

SECONDARY OUTCOMES:
Postpaortum period- Post-discharge | Post-discharge - one month after birth
  Evaluation of incontinence score with the Michigan Incontinence Severity Index Form( minimum score: 0 - maximum score: 40; seven and above was accepted as the cut-off point) after discharge, after one month of childbirth. Questions 1st-3th on the Michigan Incontinence Severity Index Form indicate stress incontinence severity, 4th-6th questions measure the severity of urge incontinence, and 1st-8th questions measure the severity of incontinence. There points and above indicate stress incontinence and the total score of questions 4-6 indicates 5 points and above for urge incontinence severity.A score higher than the given cut-off values indicates that the severity of incontinence is worsening.

OTHER OUTCOMES:
Birth Outcomes | After labor in 48 hour
  To evaluate the effect of prenatal pilates-assisted birth preparation training on the duration of birth (hours, minutes), the analgesia/anesthesia used, and the mode of birth rate (number and percentage) with the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Buran, Asis Prof, Principal Investigator — Uludag University
Locations (1):
- Bursa Uludağ Üniversitesi, Nilufer, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Mazzarino M, Kerr D, Morris ME. Pilates program design and health benefits for pregnant women: A practitioners' survey. J Bodyw Mov Ther. 2018 Apr;22(2):411-417. doi: 10.1016/j.jbmt.2017.05.015. Epub 2017 May 31. PMID 29861243
- [Background] Sargin MA, Yassa M, Taymur BD, Ergun E, Akca G, Tug N. Adaptation and validation of the Michigan Incontinence Severity Index in a Turkish population. Patient Prefer Adherence. 2016 May 26;10:929-35. doi: 10.2147/PPA.S106209. eCollection 2016. PMID 27307713
- [Result] Ahlund S, Rothstein E, Radestad I, Zwedberg S, Lindgren H. Urinary incontinence after uncomplicated spontaneous vaginal birth in primiparous women during the first year after birth. Int Urogynecol J. 2020 Jul;31(7):1409-1416. doi: 10.1007/s00192-019-03975-0. Epub 2019 May 28. PMID 31139858
- [Result] Chang SR, Lin WA, Chang TC, Lin HH, Lee CN, Lin MI. Risk factors for stress and urge urinary incontinence during pregnancy and the first year postpartum: a prospective longitudinal study. Int Urogynecol J. 2021 Sep;32(9):2455-2464. doi: 10.1007/s00192-021-04788-w. Epub 2021 Apr 9. PMID 33835213
- [Result] Dias NT, Ferreira LR, Fernandes MG, Resende APM, Pereira-Baldon VS. A Pilates exercise program with pelvic floor muscle contraction: Is it effective for pregnant women? A randomized controlled trial. Neurourol Urodyn. 2018 Jan;37(1):379-384. doi: 10.1002/nau.23308. Epub 2017 May 23. PMID 28543751
- [Derived] Buran G, Erim Avci S. The effect of pregnancy pilates-assisted childbirth preparation training on urinary incontinence and birth outcomes: a randomized-controlled study. Arch Gynecol Obstet. 2024 Nov;310(5):2725-2735. doi: 10.1007/s00404-024-07653-5. Epub 2024 Jul 31. PMID 39083052